CLINICAL TRIAL: NCT05801978
Title: Systems Biological Assessment of the Durability of Vaccine Responses
Brief Title: Durability of Vaccine Responses
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency); Open Philanthropy (Other)
Responsible Party: Principal Investigator, Nadine Rouphael, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00004930; #W911NF2320019 (Other Grant/Funding Number: Defense Advanced Research Project Agency)
Record Dates: First submitted 2023-03-25; First posted 2023-04-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Vaccine Response
Keywords: Durability; Immune Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- YF-17D Vaccination (Experimental): Yellow Fever Vaccine (YF-17D) vaccination: Eligible participants will be asked to read the Vaccine Information Sheet for YF-17D per the Centers for Disease Control and Prevention (CDC) guidelines. Participants will then receive the YF-17D vaccine. They will be observed for a minimum of 20 minutes for any immediate hypersensitivity reactions. They will also be given the International Certificate of Vaccination documenting receipt of YF-17D.
  Interventions: Biological: Live Attenuated Yellow Fever 17D Vaccine
- QIV Vaccination (Experimental): Quadrivalent seasonal influenza vaccine (QIV) vaccination: Eligible participants will be asked to read the Vaccine Information Sheet for QIV per the CDC guidelines. Participants will then receive QIV. They will be observed for a minimum of 20 minutes for any immediate hypersensitivity reactions.
  Interventions: Biological: Quadrivalent seasonal influenza vaccine

INTERVENTIONS:
Biological: Live Attenuated Yellow Fever 17D Vaccine — The FDA-approved YF-17D (YF-VAX®) is a live attenuated vaccine manufactured by Sanofi Pasteur as a one-dose vial. The vaccine is prepared by culturing the 17D-204 strain of yellow fever virus, contains sorbitol and gelatin as a stabilizer, and contains no preservative. Each vial of vaccine is supplied with a separate vial of sterile diluent, which contains sodium chloride injection USP (United States Pharmacopeia) without a preservative.
  Arms: YF-17D Vaccination
Biological: Quadrivalent seasonal influenza vaccine — The FDA-approved quadrivalent seasonal influenza vaccine contains four distinct strains: two influenza A viruses and two influenza B viruses. The approved seasonal QIV will be purchased from the manufacturer to be given for each season of influenza.
  Arms: QIV Vaccination

SUMMARY:
The ability of the vaccines today to generate a long-lasting protection against infections varies greatly from one vaccine to another. The yellow fever vaccine (YF-17D) is one of the most successful vaccines ever developed, having been administered to over 600 million people globally. A single vaccination is known to induce durable protection over several decades. In contrast, the quadrivalent influenza vaccine (QIV) generates an immunity that wanes quickly with no long-lasting protection. Currently, the duration of immune protection for new vaccines is difficult to predict during vaccine product development and can only be ascertained by a "wait and see" approach. This is due, in part, to the fact that some of the signals that activate a durable immune system protection remain unknown.

This study aims to provide a better understanding of this problem by vaccinating willing participants with either the FDA-approved yellow fever vaccine or the quadrivalent influenza vaccine and collecting baseline and follow-up biologic samples to compare how the immune system reacts.

DETAILED DESCRIPTION:
The ability of the vaccines today to generate a long-lasting protection against infections varies greatly from one vaccine to another. The yellow fever vaccine (YF-17D) is one of the most successful vaccines ever developed, having been administered to over 600 million people globally. A single vaccination is known to induce durable protection over several decades. In contrast, the influenza vaccine generates an immunity that wanes quickly with no long-lasting protection. Currently, the duration of immune protection for new vaccines is difficult to predict during vaccine product development and can only be ascertained by a "wait and see" approach. This is due, in part, to the fact that some of the signals that activate a durable immune system protection remain unknown.

This study aims to provide a better understanding of this problem by vaccinating willing participants with either the FDA-approved yellow fever vaccine or the quadrivalent influenza vaccine and collecting baseline and follow-up biologic samples to compare how the immune system reacts. The biologic samples will be collected from the blood (where antibodies are), the lymph nodes (where immune cells that make antibodies are present), and from the bone marrow (where long-lived cells that secrete antibodies are found). This study will take place at the Hope Clinic of Emory University.

The participants who express interest to ads for this research will be contacted by study staff who will provide further information about the study and conduct a primary evaluation of the eligibility criteria. If the participant is interested and verifies the eligibility criteria, a screening visit will be scheduled during which the study staff will go over the informed consent form with the participant. Other study procedures will be performed during this screening visit if the participant agrees to sign the informed consent form.

This study will include a screening visit, a vaccination visit, tissue sampling visits and a series of follow-up visits. During the tissue sampling visits, one or two procedures will be performed: A) Lymph node sampling during which an expert, guided by imaging, will take fine needle aspirates/ core biopsies from a lymph node. B) Bone marrow aspirate during which an expert will aspirate a small amount of bone marrow. Lymph node sampling procedures will be performed no more than two times each and bone marrow aspirations will be performed no more than three times each on the same participant. Other study procedures include a collection of medical history and medications taken, a urine pregnancy test for participants who are biologically able to become pregnant, a recording of vital signs, and a collection of adverse events that the participant experiences during their participation in the study. An HIV test is obtained as well at screening. Memory Aid will be completed by each participant.

The blood, lymph node, and bone marrow samples collected during this study will be stored and tested to evaluate how the immune system has responded to the vaccination over time. The remaining unused samples will be stored for use in future research.

This research will help advance the knowledge the study team has of how the immune system reacts to different vaccines, which will in turn, enable to identification of the factors that help predict the extent of durability of protection gained from a specific vaccine. This will also have a major impact on the way future vaccines are developed to provide long-lasting immunity against infections.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and give informed consent.
* Age 18-50 years.
* Participants agree not to take any live vaccines 30 days before or after (14 days for inactivated) vaccination.
* Women of child bearing potential must agree to use effective birth control for the first 3 months of the study. A negative urine pregnancy test must be documented prior to vaccination and prior to tissue sampling procedures.

Exclusion Criteria:

* History of allergy or serious adverse reaction, including Guillain-Barré syndrome, to a vaccine or vaccine products.
* History of a medical condition resulting in impaired immunity (such as HIV infection, cancer, particularly leukemia, lymphoma, use of immunosuppressive or antineoplastic drugs or X-ray treatment). Persons with previous skin cancers or cured non-lymphatic tumors are not excluded from the study.
* History of Hepatitis B or Hepatitis C infection.
* Chronic clinically significant medical problems that could affect the immune response, require medication that would affect the immune response, or have signs or symptoms that could be confused with reactions to vaccination, including (but not limited to):

  1. Insulin dependent diabetes
  2. Severe heart disease (including arrhythmias)
  3. Severe lung disease
  4. Severe liver disease
  5. Severe kidney disease
  6. Grade 4 hypertension (*Grade 4 hypertension per CTCAE criteria is defined as life-threatening consequences (e.g., malignant hypertension, transient or permanent neurologic deficit))
* Thymus gland problems (such as myasthenia gravis, DiGeorge syndrome, thymoma) or removal of thymus gland or history of uncontrolled autoimmune disorder.
* Pregnancy or breast feeding, or plans to become pregnant in the first 3 months of study participation.
* Receipt of blood products or immune globulin product within the prior 3 months.
* Active duty military.
* History of excessive alcohol consumption, drug use, psychiatric conditions, social conditions or occupational conditions that in the opinion of the investigator would preclude compliance with the trial.

Additional Exclusion Criteria for YF-17D Arm

* History of previous yellow fever, West Nile, Dengue, St. Louis encephalitis, or Japanese encephalitis vaccination or infection.
* Previous residence in a country where there is a risk of yellow fever virus (YFV) transmission
* History of allergy to eggs, chicken, or gelatin.

Additional Exclusion Criteria for QIV Arm

* History of influenza infection within the same influenza season.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Magnitude of neutralizing antibody (nAB) response against YF-17D in blood | Up to 270 days after vaccination
  Magnitude of neutralizing antibody responses against YF-17D at 270 days after vaccination among participants who receive YF-17D.
Magnitude of neutralizing antibody (nAb) response against QIV in blood | Up to 270 days after vaccination
  Magnitude of neutralizing antibody responses against influenza vaccine strains at 270 days after vaccination among participants who receive QIV.

SECONDARY OUTCOMES:
Frequency of adverse events until day 28 | Until day 28 after vaccination with YF-17D or QIV
  Adverse events of grade 2 or higher (AE, defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of vaccine, without any judgment about causality) will be identified during questioning or examination of participants during study visits or receiving a safety contact from a participant.
Severity of adverse events until day 28 | Until day 28 after vaccination with YF-17D or QIV
  Adverse events (AE) will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0
Frequency of serious adverse events until day 270 | Until day 270 after vaccination with YF-17D or QIV
  Serious adverse events (SAE, defined as an AE that in the view of the investigator results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect) will be identified during questioning or examination of participants during study visits or receiving a safety contact from a participant any time during the study.
Severity of serious adverse events until day 270 | Until day 270 after vaccination vaccination with YF-17D or QIV
  SAE will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0.
Frequency of adverse events until day 7 after lymph node sampling and/or bone marrow aspiration | Until day 7 after lymph node sampling and/or bone marrow aspiration
  Adverse events (AE) of grade 2 or higher will be identified during questioning or examination of participants during study visits, telephone calls 7 +/- 3 days after lymph node sampling and/or bone marrow aspiration, or receiving a safety contact from a participant.
Severity of adverse events until day 7 after lymph node sampling and/or bone marrow aspiration | Until day 7 after lymph node sampling and/ or bone marrow aspiration
  SAE will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - The Hope Clinic of Emory University, Decatur, Georgia